CLINICAL TRIAL: NCT00957944
Title: Single-site, Open-label, Randomized, Cross-over Trial to Evaluate the Bioequivalence of Single Dose Rotigotine Transdermal Patch (4.5 mg/10 cm^2) From 2 Different Manufacturing Sites.
Brief Title: Study in Healthy Volunteers to Prove That Two Rotigotine Patches From Different Manufacturing Sites Deliver Equivalent Drug Amount to the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SP0957
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2010-09-22 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2012-04

CONDITIONS: Healthy Volunteers
Keywords: Rotigotine; Neupro®
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A-B (Test: PR 2.1.1 WCL - Reference: PR 2.1.1 AND) (Experimental): Two single applications of rotigotine patches from two different manufacturing sites in the order A-B separated by a washout phase of at least 5 days
  Interventions: Drug: rotigotine transdermal patch (Neupro®)
- Sequence B-A (Reference: PR 2.1.1 AND - Test: PR 2.1.1 WCL) (Experimental): Two single applications of rotigotine patches from two different manufacturing sites in the order B-A separated by a washout phase of at least 5 days
  Interventions: Drug: rotigotine transdermal patch (Neupro®)

INTERVENTIONS:
Drug: rotigotine transdermal patch (Neupro®) — Rotigotine 4.5 mg/10 cm^2 patch applied for 24 hours
  Other Names: Neupro®

SUMMARY:
The major aim of this study is to investigate and compare the drug amount delivered to the body after sequential application of 2 rotigotine transdermal patches from 2 different manufacturing sites.

ELIGIBILITY:
Inclusion Criteria:

* healthy, white, male volunteers between 18 and 55 years of age (inclusive)
* BMI between 19 and 28 kg/m² (inclusive)

Exclusion Criteria:

* previous participation in a clinical study with Rotigotine
* history or current condition of epilepsy and/or seizures
* known clinically relevant allergy or known/suspected clinically relevant drug hypersensitivity
* history of significant skin hypersensitivity to adhesives or other transdermal products or recently unresolved contact dermatitis
* history or present condition of an atopic or eczematous dermatitis, psoriasis, and/or an active skin disease
* clinically relevant abnormality in physical examination, ECG, vital signs or safety laboratory examinations
* positive HIV, hepatitis B or C test or positive alcohol or drug test
* relevant hepatic or renal dysfunction
* intake of medication that might interfere with the test drug within 2 weeks prior to dosing
* thickly hair-covered abdomen resulting in difficulties in finding appropriate patch application sites

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Neuss, North Rhine-Westphalia, Germany

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 40 healthy, male subjects has been randomized in order to complete the trial with at least 30 subjects eligible for the Pharmacokinetic Set (PKS). Baseline characteristics refer to the PKS.
Pre-assignment Details: One subject that fulfilled predefined criteria for patch adhesiveness was excluded from the PKS.
Groups:
- Sequence A-B (Test: PR 2.1.1 WCL - Reference: PR 2.1.1 AND): Treatment A (Rotigotine transdermal patch 4.5 mg/10 cm^2 manufactured at LTS West Caldwell, USA) in first intervention period and Treatment B (Rotigotine transdermal patch 4.5 mg/10 cm^2 manufactured at LTS Andernach, Germany) in second intervention period (after washout period of at least 5 days)
- Sequence B-A (Reference: PR 2.1.1 AND - Test: PR 2.1.1 WCL): Treatment B (Rotigotine transdermal patch 4.5 mg/10 cm^2 manufactured at LTS Andernach, Germany) in first intervention period and Treatment A (Rotigotine transdermal patch 4.5 mg/10 cm^2 manufactured at LTS West Caldwell, USA) in second intervention period (after washout period of at least 5 days)
Period: First Intervention- 24 Hours
Arm/Group | Sequence A-B (Test: PR 2.1.1 WCL - Reference: PR 2.1.1 AND) | Sequence B-A (Reference: PR 2.1.1 AND - Test: PR 2.1.1 WCL)
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout Period of at Least 5 Days
Arm/Group | Sequence A-B (Test: PR 2.1.1 WCL - Reference: PR 2.1.1 AND) | Sequence B-A (Reference: PR 2.1.1 AND - Test: PR 2.1.1 WCL)
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0
Period: Second Intervention- 24 Hours
Arm/Group | Sequence A-B (Test: PR 2.1.1 WCL - Reference: PR 2.1.1 AND) | Sequence B-A (Reference: PR 2.1.1 AND - Test: PR 2.1.1 WCL)
Started | 20 | 19
Pharmacokinetic Set (PKS) | 20 | 18 (One subject that fullfilled predefined criteria for patch adhesiveness was excluded from the PKS)
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A-B (Test: PR 2.1.1 WCL - Reference: PR 2.1.1 AND) | Sequence B-A (Reference: PR 2.1.1 AND - Test: PR 2.1.1 WCL) | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (11.7) | 32.8 (7.2) | 35.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 18 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 18 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 18 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI= Weight/(Height)^2
  kilogram per square meter (kg/m^2) | 25.03 (2.16) | 25.87 (1.77) | 25.43 (2.00)
Height [Mean (Standard Deviation); unit: meter (m)] | 1.82 (0.07) | 1.82 (0.08) | 1.82 (0.08)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 83.18 (9.62) | 85.33 (8.75) | 84.20 (9.16)

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-tz) of Unconjugated Rotigotine
Description: The AUC(0-tz) is the area under the plasma concentration- time curve from zero up to the last analytically quantifiable concentration.
Time Frame: Pharmacokinetic samples were taken predose, after 1, 2, 3, 4, 6, 8, 12, 16, 24 (before patch removal), 25, 26, 28, 30, 32, 36, 40 and 48 hours after patch application.
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: (ng/ mL)*h
Groups:
- Treatment A (Test: PR 2.1.1 WCL): Rotigotine transdermal patch (4.5 mg/10 cm^2) manufactured at LTS West Caldwell, USA (Test; drug product PR2.1.1 WCL); single application of 1 patch for 24 hours
- Treatment B (Reference: PR 2.1.1 AND): Rotigotine transdermal patch (4.5 mg/10 cm^2) manufactured at LTS Andernach, Germany (Reference; drug product PR2.1.1 AND); single application of 1 patch for 24 hours
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
(ng/ mL)*h | 4.3899 (1.7959) | 4.4255 (2.3969)
Statistical Analysis 1: Comparison: Treatment A (Test: PR 2.1.1 WCL) vs Treatment B (Reference: PR 2.1.1 AND); Bioequivalence testing by using the 90% Confidence Interval (CI); Test type: Non-Inferiority or Equivalence — If the 90% Confidence Interval for the ratio of geometric LS- Means is included within 0.8- 1.25, the patches are considered bioequivalent; ANOVA; ANOVA for log- transformed values has been used as the basis for calculation of point estimates (LS- Means) and Confidence Intervals (CIs); ratio of geometric LS- Means = 1.0302, 90% CI [0.9693 to 1.0951] — Bioequivalence is concluded if the 90% CIs for the ratio Treatment A/ Treatment B are fully included in the acceptance range from 0.8- 1.25 for AUC(0-tz), AUC(0-inf) and Cmax

2. Primary Outcome: Cmax of Unconjugated Rotigotine
Description: The Cmax is the maximum plasma concentration.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: ng/ mL
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
ng/ mL | 0.21103 (0.08827) | 0.20386 (0.10194)
Statistical Analysis 1: Comparison: Treatment A (Test: PR 2.1.1 WCL) vs Treatment B (Reference: PR 2.1.1 AND); Bioequivalence testing by using the 90% Confidence Interval (CI); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; ratio of geometric LS- Means = 1.0571, 90% CI [0.9903 to 1.1284] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC(0-∞) of Unconjugated Rotigotine
Description: The AUC(0-∞) is the area under the plasma concentration- time curve from zero up to infinity
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: (ng/ mL)*h
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
(ng/ mL)*h | 4.51237 (1.80709) | 4.55159 (2.42524)
Statistical Analysis 1: Comparison: Treatment A (Test: PR 2.1.1 WCL) vs Treatment B (Reference: PR 2.1.1 AND); Bioequivalence testing by using the 90% Confidence Interval (CI); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; ratio of geometric LS- Means = 1.0289, 90% CI [0.9714 to 1.0899] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: AUC(0-tz) Norm (Apparent Dose) of Unconjugated Rotigotine
Description: The AUC(0-tz) norm (apparent dose) is the area under the plasma concentration- time curve from zero up to the last analytically quantifiable concentration normalized by apparent dose (mg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: (ng/ mL)*(h/ mg)
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
(ng/ mL)*(h/ mg) | 2.23980 (0.71015) | 2.23035 (0.77992)

5. Secondary Outcome: AUC(0-tz) Norm (BW) of Unconjugated Rotigotine
Description: The AUC(0-tz) norm (BW) is the area under the plasma concentration- time curve from zero up to the last analytically quantifiable concentration normalized by body weight (kg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: (ng/ mL)*h*kg
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
(ng/ mL)*h*kg | 364.930 (140.747) | 367.452 (189.279)

6. Secondary Outcome: AUC(0-∞) Norm (Apparent Dose)
Description: The AUC(0-∞) norm (apparent dose) is the area under the plasma concentration- time curve from zero up to infinity normalized by apparent dose (mg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: (ng/ mL)*(h/ mg)
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
(ng/ mL)*(h/ mg) | 2.30523 (0.71105) | 2.29747 (0.78191)

7. Secondary Outcome: AUC(0-∞) Norm (BW)
Description: The AUC(0-∞) norm (BW) is the area under the plasma concentration- time curve from zero up to infinity normalized by body weight (kg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: (ng/ mL)*h*kg
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
(ng/ mL)*h*kg | 375.224 (141.465) | 378.003 (191.344)

8. Secondary Outcome: Cmax,Norm (Apparent Dose) of Unconjugated Rotigotine
Description: The Cmax,norm (apparent dose) is the maximum plasma concentration normalized by apparent dose(mg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: (ng/ mL)/ mg
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
(ng/ mL)/ mg | 0.108148 (0.037618) | 0.103965 (0.035474)

9. Secondary Outcome: Cmax,Norm (BW) of Unconjugated Rotigotine
Description: The Cmax,norm (BW) is the maximum plasma concentration normalized by body weight(kg).
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: (ng/ mL) * kg
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
(ng/ mL) * kg | 17.6070 (7.2645) | 16.9748 (8.1930)

10. Secondary Outcome: Tmax of Unconjugated Rotigotine
Description: The tmax is the time to reach a maximum plasma concentration after patch application.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
hour (h) | 16.00 (4.92) [8.00 to 25.00] | 16.00 (5.12) [8.00 to 26.00]

11. Secondary Outcome: MRT of Unconjugated Rotigotine
Description: The MRT is the mean residence time.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
hour (h) | 19.914 (1.620) | 19.980 (2.038)

12. Secondary Outcome: λz of Unconjugated Rotigotine
Description: The λz is the rate constant of elimination.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: 1/ hour (1/h)
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
1/ hour (1/h) | 0.129745 (0.026292) | 0.125217 (0.027732)

13. Secondary Outcome: t1/2 of Unconjugated Rotigotine
Description: The t1/2 is the terminal half- life.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
hour (h) | 5.5408 (1.0205) | 5.7878 (1.1985)

14. Secondary Outcome: CL/f of Unconjugated Rotigotine
Description: The CL/f is the apparent total body clearance.
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
L/h | 1185.98 (574.45) | 1227.56 (541.82)

15. Secondary Outcome: Apparent Dose
Description: Apparent dose of unconjugated rotigotine in mg. The apparent dose of unconjugated rotigotine was determined from the patches removed on Day 2.
Time Frame: 48 hours
Population: Pharmacokinetic Set (PKS)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Number analyzed (Participants) | 38 | 38
mg | 1.932 (0.398) | 1.927 (0.489)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected up to 18 days from Day -1 (day before first dosing) to the Safety Follow- Up Visit.
Description: Adverse Events (AEs) refer to the Safety Set (SS). The SS includes all subjects who are randomized and received at least one dose of study medication.
Arm/Group | Treatment A (Test: PR 2.1.1 WCL) | Treatment B (Reference: PR 2.1.1 AND)
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 5/39 | 6/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (Test: PR 2.1.1 WCL) (N=39) | Treatment B (Reference: PR 2.1.1 AND) (N=40)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Application Site Pruritus (General disorders) | 4 (4) | 3 (3)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Sleep Disorder (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.